CLINICAL TRIAL: NCT01817504
Title: Interest of Systematic Transplantectomy Versus Conventional Care After Kidney Graft Failure
Brief Title: Systematic Transplantectomy Versus Conventional Care After Kidney Graft Failure
Acronym: DESYRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012.714; 2012-A00421-42 (Other: ANSM)
Record Dates: First submitted 2013-03-08; First posted 2013-03-25 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Renal Transplantation
Keywords: Renal failure,; Transplantectomy; Immunosuppression; Sensitization
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): The study group corresponds to systematic transplantectomy under immunosuppressive therapy within two months after return to dialysis,
  Interventions: Procedure: Systematic transplantectomy
- Control group (Other): The control group corresponds to progressive reduction of immunosuppression without systematic transplantectomy after return to dialysis
  Interventions: Procedure: Progressive reduction of immunosuppression

INTERVENTIONS:
Procedure: Systematic transplantectomy — Transplantectomy within two months after return to dialyse. Antiproliferatives stop at the start of dialysis. Maintenance basic immunosuppressive treatment without dose reduction up to two weeks after transplantectomy. Abrupt discontinuation of the basic immunosuppressive treatment ttwo weeks after transplantectomy. Maintenance corticosteroids at 5mg per day until one month after transplantectomy then stop corticosteroids within one month.
  Arms: Study group
Procedure: Progressive reduction of immunosuppression — Progressive reduction of immunosuppression. Transplantectomy for cause only. Antiproliferatives withdrawn at the start of dialysis. Maintenance of anticalcineurin or mTOR inhibitors half dose for 3 months, ¼ dose for 3 months and then stop. Maintenance corticosteroids for 6 months up to 5 mg per day, and then soft stop in 3 months.
  In case of transplantectomy by reason in the control group, basic immunosuppression will be continued at the maintenance dose during the current surgical procedure, and withdrawn two weeks later, similary to the strategy used in the study group.
  Arms: Control group

SUMMARY:
Our hypothesis is early and systematic transplantectomy under a well-conducted immunosuppression is associated with a decreased risk of anti-HLA immunization against a conservative attitude including a gradual reduction of immunosuppression, with or without a transplantectomy performed for cause (clinical event).

Observation or Investigation Method Used :

The study is :

* multicenter
* prospective
* open
* randomized: patients are divided into two parallel groups:

  * study group: transplantectomy within six weeks after return to dialysis, antiproliferatives stop at the start of dialysis, Maintenance anticalcineurin-based-immunosuppression without dose reduction up to two weeks after transplantectomy. Abrupt discontinuation of anticalcineurin two weeks after transplantectomy. Corticosteroids: 5mg per day until one month after transplantectomy then stop within one month.
  * control group: No systematic transplantectomy. Antiproliferatives stop at the start of dialysis.Anticalcineurins half dose for 3 months, ¼ dose for 3 months and then stop. Corticosteroids:5 mg per day for 6 months, and then tapered and stop within 3 months.

In the case of transplantectomy for cause in the control group, immunosuppression will be continued at the maintenance dose during the current surgical procedure, and withdrawn two weeks later,similary to systematic transplantectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years.
* Patients affiliated to health protection system, social security in France or any similar regimen.
* Renal transplant patient with end-stage transplantation, regardless of the number of previous transplants.
* Patient receiving immunosuppressive protocol based on anticalcineurin or mTOR inhibitors
* Patient should have resume hemodialysis within 4 weeks
* Duration of transplantation more than one year
* Patient with asymptomatic graft
* immunogenic potential residual >50% (calculated PIR during the re-dialysis)
* Patient not covered by any measure of legal protection.

Exclusion Criteria:

* Immunogenic potential residual <50%
* Graft infection uncontrolled by treatment
* Active infectious pathology
* Inflammatory graft
* Uncontrolled arterial hypertention
* Inflammatory syndrome of undetermined origin with CRP>50mg/l
* Fever of unknown origin for more than 8 days T>38°C
* Contra-indication to surgery
* AVK treatment
* Patient candidate for a living donor within 12 months
* Monotherapy with calcineurin inhibitors or mTOR inhibitors
* Treatment directed against the humoral response in the 6 months preceding the recovery of dialysis (Rituximab IV-Ig or high doses)
* Presence of another transplant (pancreas, liver, heart, lung)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Anti HLA Immunization assessed by Luminex assay | 12 months (M12)
  Evaluate the interest of a transplantectomy early (<2 months after return to dialysis) and systematic under immunosuppressive in renal transplant patients after loss of renal graft function in terms of anti-HLA immunization (measured by Luminex test) a year after loss of renal graft function and return to dialysis in the renal transplant patient.
  Proportion of patients who developed HLA immunization (DSA)after systematic transplantectomy under immunosuppression versus progressive reduction of immunosuppression without transplantectomy

SECONDARY OUTCOMES:
Kinetics anti-HLA antibodies after transplantectomy | 12 months after inclusion
  Determine the kinetics of new onset anti-HLA antibodies at D0, D15, D30, M3, M6, M9 after systematic or for cause transplantectomy and in the year following graft failure and the proportion of immunized patients during the first 6 months after dialysis. HLA antibodies will be assessed by Luminex test. The specificity of antibodies against HLA I or HLA II will be determined, as well as Mean Immunofluorescence Intensity in each case.
Morbidity and mortality after transplantectomy | 12 months after inclusion
  Determine the morbidity and mortality after transplantectomy according to its indication, systematic or for cause (transplantectomy indications in the control group: persistent pain graft, unexplained fever, hematuria, inflammation or unexplained anemia ).
Measuring the impact of systematic transplantectomy on mortality, inflammation, nutritional status, anemia, hypertension and cardiovascular risk factors | 12 months
  The following parameters will be measured at D0, M1, M3, M6, M9 and M12 after return to dialysis during the first year after kidney graft failure: CRP, pre-albuminemia, albuminemia, BMI, hemoglobin, hematocrit, blood pressure, cholesterol, LDL cholesterol and triglyceride.
Infectious comorbidity | 12 months
  The impact of early cessation of immunosuppression on infectious complications after kidney graft failure will assessed. For each patient, origin of infection, bacterial, viral, fungal, will determined. The total number of infection episodes during the first year will be analyzed in the two groups.
Costs of two strategies | 12 months after inclusion
  To evaluate the medico-economic impact of each conservation strategy in the management of patients who return to dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MORELON, MD, Principal Investigator — Transplantation Department, Hopital Edouard Herriot, Hospices Civils de Lyon
Locations (9):
- France (9):
  - Service de Néphrologie et Transplantation Rénale, CHU Gabriel Montpied, Clermont-Ferrand
  - Service de Néphrologie -Dialyse-Transplantation, Hôpital Michallon, Grenoble
  - Transplantation Department, Hôpital Edourad Herriot, Lyon
  - Service de Néphrologie et Transplantation Rénale - Hôpital Lapeyronie, Montpellier
  - Institut de Transplantation, Urologie et Néphrologie - CHU Nantes, Nantes
  - Service de Néphrologie-Dialyse, Centre Hospitalier d'Annecy, Pringy
  - Service de Néphrologie, Dialyse et Transplantation Rénale, Hôpital Nord, Saint-Etienne
  - Service de Néphrologie et Transplantation Rénale - Nouvel Hôpital Civil, Strasbourg
  - Service de Néphrologie, Immunologie Clinique - CHU Bretonneau, Tours